CLINICAL TRIAL: NCT02433379
Title: Understanding Outcomes With the EMBLEM™ S-ICD in Primary Prevention Patients With Low Ejection Fraction
Acronym: UNTOUCHED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 91026550
Record Dates: First submitted 2015-04-23; First posted 2015-05-05 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia; Low Cardiac Output
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Cardiac Output, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Subjects implanted with an EMBLEM S-ICD with rate zones set at 200 bpm and 250 bpm per protocol.
  Interventions: Device: EMBLEM S-ICD System

INTERVENTIONS:
Device: EMBLEM S-ICD System — The intervention comprises programming the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) with zone cutoffs at 200 bpm and 250 bmp

SUMMARY:
This study assesses the 18-month incidence of inappropriate shocks in subjects implanted with the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) for primary prevention of sudden cardiac death. Devices are to be programmed with zone cutoffs at 200 bpm and 250 bmp in order to mimic the programming settings for transvenous ICDs in the MADIT RIT study. The incidence of inappropriate S-ICD shocks will be compared to the incidence of inappropriate shocks observed in the MADIT RIT study.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillator (ICD) therapy is highly effective for reducing mortality in patients with clinical markers for elevated risk for ventricular arrhythmias. However, inappropriate shocks and unnecessary appropriate shocks remain an important side effect that can significantly affect an ICD recipient's quality of life and may be deleterious to the myocardium.

The MADIT RIT study demonstrated that the incidence of inappropriate and unnecessary appropriate ICD therapy can be reduced in primary prevention patients through two different programming strategies: 1) High Rate Zone Cutoff, i.e., raising the lowest rate detection cutoff to 200 bpm; and 2) Delayed Therapy Initiation, i.e., increasing the time to therapy initiation to 60 seconds for arrhythmias detected between 170-199 bpm and 12.5 seconds between 200-249 bpm. Both strategies effectively reduced the amount of ICD therapy delivered when compared to conventional programming, where the lowest rate detection cutoff was 170 bpm and the delay to therapy initiation was programmed to 2.5 seconds. Importantly, neither treatment arm was associated with significantly increased syncope or mortality. The results of MADIT RIT established preferred device settings for reducing shocks in transvenous ICD (TV-ICD) patients with a primary prevention indication.

Preferred settings for subcutaneous ICDs, however, have not been established with data from prospective studies. The UNTOUCHED study will test a programming scheme designed to minimize inappropriate and unnecessary shocks in patients who have an indication for primary prevention of sudden cardiac death and low ejection fraction. Although S-ICD programming options do not permit exact replication of the programmed settings previously shown to reduce shocks in the MADIT RIT treatment arms, key elements are combined into the UNTOUCHED settings to be tested in this protocol. It is hypothesized that despite the lack of anti-tachycardia pacing, the EMBLEM S-ICD settings utilized in this study will result in an overall shock incidence similar to that observed in ICD patients from MADIT RIT.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ischemic or non-ischemic heart disease who meets current guidelines for ICD therapy and intends to undergo a de novo implant procedure for an EMBLEM™ S-ICD (or newer generation BSC S-ICD)
* Left ventricular ejection fraction ≤ 35%
* A passing EMBLEM™ S-ICD (or newer generation BSC S-ICD) screening ECG
* Patient ≥ 21 years of age willing and capable of giving informed consent
* Patient willing and capable of complying with follow-up visits

Exclusion Criteria:

* Patient with a history of spontaneous sustained VT or VF
* Patient with bradycardia pacing indication
* Patient eligible and scheduled for cardiac resynchronization implant
* Patient with a previous S-ICD or a previous transvenous pulse generator (pacemaker or defibrillator)
* Patient in NYHA Class IV documented in the medical records within 90 days before enrollment
* Patient with life expectancy shorter than 18 months due to any medical condition (e.g., cancer, uremia, liver failure, etc…)
* Patient receiving hemodialysis within 180 days before to enrollment
* Patients unable to give consent in person, including patients unable to read or write
* Patient who is known to be pregnant or plans to become pregnant over the course of the trial
* Patient unwilling or unable to cooperate with the protocol
* Participation in concurrent clinical study without prior approval from Boston Scientific
* Medical status (e.g., hemodynamic conditions ) of the patient doesn't allow programming devices with a conditional shock zone at 200 bpm and a shock zone at 250 bpm, in the judgment of the implanting physician and/or according to (inter) national guidelines

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, Principal Investigator — Medical University of South Carolina; Lucas Boersma, MD, Principal Investigator — St. Antonius Hospital
Locations (110):
- United States (69):
  - Alabama Cardiovascular Group, Birmingham, Alabama
  - Huntsville Hospital - The Heart Center, PC, Huntsville, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Glendale Adventist Medical Center, Glendale, California
  - Sharp Grossmont Hospital, La Mesa, California
  - University of Southern California Hospital, Los Angeles, California
  - Alta Bates Medical Center, Oakland, California
  - St. Joseph Hospital, Orange, California
  - Good Samaritan Hospital - San Jose, San Jose, California
  - Harbor UCLA Medical Center, Torrance, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Cardiology Physicians PA, Newark, Delaware
  - Baptist Medical Center, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - CorVita Science Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northern Indiana Research Alliance - Lutheran Hospital, Fort Wayne, Indiana
  - Methodist Hospital of Indianapolis, Indianapolis, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Heartland Cardiology, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CardioVascular Institute of Michigan P.C., Roseville, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Mercy Research, Springfield, Missouri
  - Cox Health, Springfield, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - HealthCare Partners Cardiology, Las Vegas, Nevada
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cooper Hospital - University Medical Center, Camden, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - Albany Medical Center, Albany, New York
  - Northwell Health, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Salem Hospital, Salem, Oregon
  - Sacred Heart Medical Center at Riverbend, Springfield, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Centra Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - CHI Franciscan Health System, Tacoma, Washington
  - St. Mary's Madison, Madison, Wisconsin
- Belgium (2):
  - Clinique Saint-Jean, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Institut universitaire de Cardiologie et de Pneumologie de Quebec, Ste-Foy, Quebec, Canada
- University Hospital, Odense, Denmark
- France (10):
  - CH Annecy, Annecy
  - CHU Dijon, Dijon
  - CHRU de Lille, Lille
  - CHU La Timone Hospital, Marseille
  - CHU Montpellier, Montpellier
  - Hospital de la Pitie-Salpetriere, Paris
  - CHRU Hopital Pontchaillou, Rennes
  - Nouvel Hôpital Civil De Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Unfallkrankenhaus Berlin Marzahn, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - University Hospital Frankfurt, Frankfurt
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitaetsklinik Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University Hospital of Muenster, Münster
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC - University Medical Center Rotterdam, Rotterdam
- Centralny Szpital Kliniczny Uniwerytetu Medycznego, Lodz, Poland
- Hospital San Lucas, Ponce, Puerto Rico
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen De La Salud, Toledo
  - Hospital Miguel Servet, Zaragoza
- Switzerland (2):
  - Cardiocentro Ticino, Lugano
  - University Hospital Zurich, Zurich
- United Kingdom (7):
  - Blackpool Victoria NHS Trust Direct, Blackpool
  - Russels Hall Hospital, Dudley
  - Glenfield Hospital, Leicester
  - Cardiothoracic Centre, Liverpool
  - St. Bartholomews Hospital, London
  - Northern General Hospital, Sheffield
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066
- [Background] Gold MR, Knops R, Burke MC, Lambiase PD, Russo AM, Bongiorni MG, Deharo JC, Aasbo J, El Chami MF, Husby M, Carter N, Boersma L. The Design of the Understanding Outcomes with the S-ICD in Primary Prevention Patients with Low EF Study (UNTOUCHED). Pacing Clin Electrophysiol. 2017 Jan;40(1):1-8. doi: 10.1111/pace.12994. Epub 2017 Jan 15. PMID 27943348
- [Result] Boersma LV, El-Chami MF, Bongiorni MG, Burke MC, Knops RE, Aasbo JD, Lambiase PD, Deharo JC, Russo AM, Dinerman J, Shaik N, Barr CS, Carter N, Appl U, Brisben AJ, Stein KM, Gold MR. Understanding Outcomes with the EMBLEM S-ICD in Primary Prevention Patients with Low EF Study (UNTOUCHED): Clinical characteristics and perioperative results. Heart Rhythm. 2019 Nov;16(11):1636-1644. doi: 10.1016/j.hrthm.2019.04.048. Epub 2019 May 10. PMID 31082539
- [Result] Gold MR, Lambiase PD, El-Chami MF, Knops RE, Aasbo JD, Bongiorni MG, Russo AM, Deharo JC, Burke MC, Dinerman J, Barr CS, Shaik N, Carter N, Stoltz T, Stein KM, Brisben AJ, Boersma LVA; UNTOUCHED Investigators*. Primary Results From the Understanding Outcomes With the S-ICD in Primary Prevention Patients With Low Ejection Fraction (UNTOUCHED) Trial. Circulation. 2021 Jan 5;143(1):7-17. doi: 10.1161/CIRCULATIONAHA.120.048728. Epub 2020 Oct 19. PMID 33073614

RESULTS

PARTICIPANT FLOW:
Groups:
- UNTOUCHED Study Participants: There were 1173 patients who were consented for participation in the UNTOUCHED Study. Of the 1173 participants enrolled 1116 were implanted or attempted for implant with an EMBLEM S-ICD and programmed with rate zones set at 200 bpm and 250 bpm per protocol. There were 57 enrolled subjects who were determined to be screen failures or were not attempted for implant. These subjects were not followed for the study and therefore not included in the study analyses/results.
Period: Overall Study
Arm/Group | UNTOUCHED Study Participants
Started | 1173
Completed | 852
Not Completed | 321
Not completed — Screen Failures | 55
Not completed — Death | 57
Not completed — Total Withdrawals | 209

BASELINE CHARACTERISTICS:
Population: UNTOUCHED Study subjects who were implanted or attempted for implant are included in the Baseline Demographics.
Groups:
- UNTOUCHED Implanted/Attempted Subjects: UNTOUCHED Study subjects who were implanted or attempted for implant with an EMBLEM S-ICD with rate zones set at 200 bpm and 250 bpm per protocol.
  EMBLEM S-ICD System: The intervention comprises programming the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) with zone cutoffs at 200 bpm and 250 bmp.
Arm/Group | UNTOUCHED Implanted/Attempted Subjects
Number analyzed (Participants) | 1116
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286
  Male | 830
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 704
  Black | 239
  Hispanic or Latino | 53
  Asian | 20
  Pacific Islander | 3
  Native American | 6
  Other | 8
  Unknown | 83
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 1
  United States | 807
  Europe | 292
  Canada | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Did Not Experience an Inappropriate Shock From Their EMBLEM S-ICD
Description: Primary endpoint: Inappropriate shock free rate from 0 to 540 Days (18-Months) compared to a performance goal of 91.6%.
Time Frame: 18 months
Population: All implanted subjects were included in the analysis except for one participant who was co-enrolled in another study that may have affected the results of this analysis. There were 4 subjects who were attempted to be implanted but did not receive a device and therefore not included in the analysis. The endpoint was analyzes using intent to treat analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- S-ICD: Subjects implanted with an EMBLEM S-ICD with rate zones set at 200 bpm and 250 bpm per protocol.
  EMBLEM S-ICD System: The intervention comprises programming the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) with zone cutoffs at 200 bpm and 250 bmp
Arm/Group | S-ICD
Number analyzed (Participants) | 1111
Percentage of participants | 95.9 [94.8 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

2. Secondary Outcome: Percentage of Participants Not Experiencing a System or Procedure Related Complication From 0 to 30 Days
Description: Secondary safety endpoint: Freedom from System and Procedure Related Complications at 30 days compared to a performance goal of 93.8%.
Time Frame: 30 days
Population: All implanted and attempted subjects were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | S-ICD
Number analyzed (Participants) | 1116
Percentage of participants | 95.8 [94.7 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

3. Secondary Outcome: Percentage of Subjects Free From All-cause Shock From Their EMBLEM S-ICD
Description: Secondary efficacy endpoint: All-Cause Shock Free Rate at 540 days (18-months) compared to a performance goal of 85.8%.
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | S-ICD
Number analyzed (Participants) | 1111
Percentage of participants | 90.6 [89.0 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

4. Other Pre Specified Outcome: Percentage of Patients Not Experiencing a System or Procedure Related Complication From 0 to 180 Days (6 Months).
Description: Post-Market Clinical Follow-up (PMCF) Endpoint: Freedom from System and Procedure Related Complications at 180 days (6 months) compared to a performance goal of 85%. This analysis was conducted for two sub-groups of UNTOUCHED Study subjects: 1.) the first 200 subjects implanted with an EMBLEM model A209 device; 2.) the first 200 subjects implanted with an EMBLEM model A219 device. The PMCF analysis prespecified in the study protocol only required a sub-set of the implanted UNTOUCHED Study subjects (i.e., 200 subjects for the EMBLEM A209 analysis and 200 for the EMBLEM A219 analysis; the full study cohort was not required for these two analyses).
Time Frame: 6 months
Population: The first 200 UNTOUCHED Study subjects implanted with an EMBLEM model A209 device as well as the first 200 UNTOUCHED Study subjects implanted with an EMBLEM model A219 device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- S-ICD (EMBLEM Model A209): The first 200 subjects implanted with an EMBLEM S-ICD (Model A209) S-ICD with rate zones set at 200 bpm and 250 bpm per protocol.
  EMBLEM S-ICD System: The intervention comprises programming the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) with zone cutoffs at 200 bpm and 250 bmp
- S-ICD (EMBLEM Model A219): The first 200 subjects implanted with an EMBLEM S-ICD (Model A219) S-ICD with rate zones set at 200 bpm and 250 bpm per protocol.
  EMBLEM S-ICD System: The intervention comprises programming the EMBLEM Subcutaneous Implantable Defibrillator (S-ICD) with zone cutoffs at 200 bpm and 250 bmp
Arm/Group | S-ICD (EMBLEM Model A209) | S-ICD (EMBLEM Model A219)
Number analyzed (Participants) | 200 | 200
Percentage of participants | 93.5 [89.9 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing). | 93.5 [89.9 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment until subjects ended their participation in the study. Subjects were considered to have completed the study after 18-Months of follow-up.
Arm/Group | S-ICD
All-Cause Mortality (participants affected / at risk) | 57/1116
Serious Adverse Events (participants affected / at risk) | 354/1116
Other Adverse Events (participants affected / at risk) | 155/1116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-ICD (N=1116)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abnormal laboratory values (Blood and lymphatic system disorders) | 4
Adverse drug reaction (General disorders) | 1
Adverse reaction - Allergic reaction (Immune system disorders) | 1
Adverse reaction - Medication (General disorders) | 1
Adverse reaction Hypotension Procedure (Injury, poisoning and procedural complications) | 3
Adverse reaction Medication/Anaphylactic shock Procedure (Injury, poisoning and procedural complications) | 2
Adverse reaction Respiratory Procedure (Injury, poisoning and procedural complications) | 5
Alcohol abuse (Psychiatric disorders) | 1
Atrial Fibrillation (AF) (Cardiac disorders) | 17
Atrial Flutter (Cardiac disorders) | 3
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 2
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 13
Cancer (General disorders) | 7
Cardiac arrest (Cardiac disorders) | 9
Cardiogenic shock (Cardiac disorders) | 12
Cerebrovascular Accident (CVA) - hemorrhagic (Vascular disorders) | 1
Cerebrovascular Accident (CVA) - ischemic (Vascular disorders) | 1
Cerebrovascular Accident (CVA) - unspecifed (Vascular disorders) | 13
Chest pain - Heart failure (Cardiac disorders) | 25
Chest pain - Ischemic (Vascular disorders) | 8
Chest pain - Other (General disorders) | 4
Coronary Artery Disease (Vascular disorders) | 17
Death (General disorders) | 10
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1
Device shocked 5 times before conversion (Product Issues) | 1
Device system discomfort (> 30d post implant) (Injury, poisoning and procedural complications) | 2
Device system infection (= 30d post implant with explant) (Infections and infestations) | 8
Device system infection (>30d post implant with explant) (Infections and infestations) | 4
Dislodgment - Oversensing - RV Lead (Product Issues) | 1
Distal thromboemboli (Vascular disorders) | 1
Dizziness (General disorders) | 2
Dizziness - Heart failure (Cardiac disorders) | 1
Drug related (General disorders) | 1
Dyspnea - Heart failure (Cardiac disorders) | 31
Electrode erosion (Skin and subcutaneous tissue disorders) | 1
Electrode migration/revision (Musculoskeletal and connective tissue disorders) | 2
Electrode migration/revision Procedure (Injury, poisoning and procedural complications) | 2
Electrode suture discomfort (Skin and subcutaneous tissue disorders) | 1
Endocrine (Endocrine disorders) | 12
Fascial defect closure (Musculoskeletal and connective tissue disorders) | 1
Fatigue - Heart failure (Cardiac disorders) | 2
Fatigue/Weakness (General disorders) | 1
Fever and/or Virus (Infections and infestations) | 11
Gastrointestinal (Gastrointestinal disorders) | 25
Genitourinary (Reproductive system and breast disorders) | 5
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 5
Heart failure symptoms - Unspecified (Cardiac disorders) | 27
Hematological (Blood and lymphatic system disorders) | 2
Hematoma - Unrelated (non study) procedure or device (Injury, poisoning and procedural complications) | 2
Hematoma PG pocket (= 30d post implant) (Injury, poisoning and procedural complications) | 4
Hemodynamic instability DFT testing Procedure (Injury, poisoning and procedural complications) | 1
Hemorrhage - Unrelated (non study) procedure or device (Injury, poisoning and procedural complications) | 3
Hypertension - Heart failure (Cardiac disorders) | 1
Hypertension/Hypertensive Crisis (Vascular disorders) | 2
Hypotension - Heart failure (Cardiac disorders) | 3
Hypotension/Orthostatic Hypotension (Vascular disorders) | 2
Hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Inadequate healing of incision site Subject (Skin and subcutaneous tissue disorders) | 1
Inadvertent arrhythmia Procedure (Injury, poisoning and procedural complications) | 2
Inappropriate tachy therapy NSC (Cardiac oversensing) Electrode (Product Issues) | 1
Inappropriate tachy therapy NSR (Cardiac oversensing) System (Product Issues) | 4
Inappropriate tachy therapy noise (Non-cardiac) System (Product Issues) | 1
Inappropriate therapy SVT above programmed rate zone System (Product Issues) | 1
Inappropriate therapy SVT discrimination error System (Product Issues) | 2
Incisional/Superficial infection (= 30d post implant without explant) (Infections and infestations) | 4
Incisional/Superficial infection (>30d post implant without explant) (Infections and infestations) | 3
Integumentary (Skin and subcutaneous tissue disorders) | 5
Intermittent ST elevation during implant (Cardiac disorders) | 1
Intracardiac thrombus (Vascular disorders) | 2
LBBB (Cardiac disorders) | 1
Localized Infection (Infections and infestations) | 7
Localized infection (Infections and infestations) | 2
Mitral regurgitation (Cardiac disorders) | 2
Multi-system failure (General disorders) | 5
Multi-system failure - Heart failure (Cardiac disorders) | 16
Multiple heart failure symptoms (Cardiac disorders) | 91
Multiple symptoms (General disorders) | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 12
Myocardial biopsy (dilated cardiomyopathy of unknown origin) (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 12
Neurological (Nervous system disorders) | 14
Non VT/VF cardiac oversensing AF (Product Issues) | 2
Out of Range shock impedance Electrode (Product Issues) | 1
Oversensing System (Product Issues) | 1
PG erosion (Skin and subcutaneous tissue disorders) | 1
PG migration Subject (Musculoskeletal and connective tissue disorders) | 1
Patient fall (Injury, poisoning and procedural complications) | 1
Peripheral edema - Heart failure (Cardiac disorders) | 1
Peripheral vascular disease (Vascular disorders) | 5
Physical trauma (Injury, poisoning and procedural complications) | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Positioning during procedure (Injury, poisoning and procedural complications) | 1
Post-surgical wound discomfort PG site (= 30d post implant) Procedure (Injury, poisoning and procedural complications) | 6
Post-surgical wound discomfort PG site (> 30d post implant) (Injury, poisoning and procedural complications) | 1
Postoperative urinary retention (Injury, poisoning and procedural complications) | 1
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1
Premature cell battery depletion - PG (Product Issues) | 3
Psychological (Psychiatric disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 21
Pulmonary Embolism (PE) (Vascular disorders) | 1
Pulmonary edema - Heart failure (Cardiac disorders) | 6
Pulseless Electrical Activity (PEA) (Cardiac disorders) | 2
Renal (Renal and urinary disorders) | 20
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Strep infection (Infections and infestations) | 1
Sub-optimal electrode position (Injury, poisoning and procedural complications) | 1
Suboptimal electrode position (Injury, poisoning and procedural complications) | 2
Suspected infection Incisional/Superficial (= 30d post implant) (Infections and infestations) | 1
Syncope (General disorders) | 1
Syncope (General disorders) | 4
Syncope - Heart failure (Cardiac disorders) | 4
Systemic infection (Infections and infestations) | 14
Transient Ischemic Attack (TIA) (Vascular disorders) | 9
Unable to convert VT/VF with S-ICD (Injury, poisoning and procedural complications) | 10
Valvular damage/Valvular insufficiency (Cardiac disorders) | 1
Vasovagal reaction (Vascular disorders) | 1
Ventricular Fibrillation (VF) (Cardiac disorders) | 4
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 12
Volume overload (Cardiac disorders) | 1
Weight gain - Heart failure (Cardiac disorders) | 4
Weight loss (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-ICD (N=1116)
AF during conversion testing (Injury, poisoning and procedural complications) | 1
Abnormal laboratory values (Blood and lymphatic system disorders) | 1
Acute blood loss (Injury, poisoning and procedural complications) | 1
Adverse reaction - General (General disorders) | 1
Adverse reaction HF symptoms Procedure (Injury, poisoning and procedural complications) | 1
Adverse reaction Hypotension Procedure (Injury, poisoning and procedural complications) | 1
Adverse reaction Medication/Anaphylactic shock Procedure (Injury, poisoning and procedural complications) | 1
Adverse reaction Respiratory Procedure (Injury, poisoning and procedural complications) | 1
Aortic stenosis (Vascular disorders) | 1
Atrial Fibrillation (AF) (Cardiac disorders) | 3
Atrial Flutter (Cardiac disorders) | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain - Heart failure (Cardiac disorders) | 21
Chest pain - Ischemic (Vascular disorders) | 1
Chest pain - Other (General disorders) | 6
Coronary Artery Disease (Vascular disorders) | 1
Dehydration - Heart failure (Cardiac disorders) | 1
Device system discomfort (> 30d post implant) (Injury, poisoning and procedural complications) | 6
Dizziness (General disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea - Heart failure (Cardiac disorders) | 3
Electrode migration/revision (Product Issues) | 1
Electrode movement Procedure (Injury, poisoning and procedural complications) | 3
Electrode suture discomfort (Injury, poisoning and procedural complications) | 1
Fatigue/Weakness (General disorders) | 1
Gastrointestinal (Gastrointestinal disorders) | 1
Genitourinary (Reproductive system and breast disorders) | 1
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1
Hematoma Electrode incision (= 30d post implant) (Injury, poisoning and procedural complications) | 1
Hematoma PG pocket (= 30d post implant) (Injury, poisoning and procedural complications) | 8
Inadequate healing of incision site Subject (Skin and subcutaneous tissue disorders) | 2
Inadvertent arrhythmia Procedure (Injury, poisoning and procedural complications) | 8
Inappropriate tachy therapy NSC (Cardiac oversensing) Electrode (Product Issues) | 2
Inappropriate tachy therapy NSR (Cardiac oversensing) System (Product Issues) | 16
Inappropriate tachy therapy noise (Non-Cardiac) PG (Product Issues) | 1
Inappropriate tachy therapy noise (Non-cardiac) System (Product Issues) | 12
Inappropriate therapy Baseline shift PG (Product Issues) | 1
Inappropriate therapy Baseline shift System (Product Issues) | 1
Inappropriate therapy SVT above programmed rate zone System (Product Issues) | 2
Inappropriate therapy SVT discrimination error System (Product Issues) | 2
Incisional/Superficial infection (= 30d post implant without explant) (Infections and infestations) | 6
Incisional/Superficial infection (>30d post implant without explant) (Infections and infestations) | 2
Incomplete header/electrode connection (Injury, poisoning and procedural complications) | 1
Integumentary (Skin and subcutaneous tissue disorders) | 1
Intermittent sensing/undersensing System (Product Issues) | 1
Multiple heart failure symptoms (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Neurological (Nervous system disorders) | 1
Non VT/VF cardiac oversensing (Product Issues) | 2
Non VT/VF cardiac oversensing AF (Product Issues) | 1
Non VT/VF cardiac oversensing for AF (Product Issues) | 1
Outcome of elective MV and LAA closure surgery (Surgical and medical procedures) | 1
Oversensing System (Product Issues) | 1
PG erosion (= 30d post implant) (Skin and subcutaneous tissue disorders) | 1
PG movement (Musculoskeletal and connective tissue disorders) | 1
Physical trauma (Injury, poisoning and procedural complications) | 2
Physical trauma Procedure (Injury, poisoning and procedural complications) | 3
Post-surgical bleeding/hemorrhage (= 30d post implant) (Injury, poisoning and procedural complications) | 1
Post-surgical wound discomfort PG site (= 30d post implant) Procedure (Injury, poisoning and procedural complications) | 20
Post-surgical wound discomfort PG site (> 30d post implant) (Skin and subcutaneous tissue disorders) | 7
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema - Heart failure (Cardiac disorders) | 1
Random component failure Therapy available System (Product Issues) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Renal (Renal and urinary disorders) | 1
Scar Cyst/Keloid Procedure (Injury, poisoning and procedural complications) | 1
Seroma PG pocket (= 30d post implant) (Injury, poisoning and procedural complications) | 1
Sinus tachycardia (Cardiac disorders) | 1
Suspected infection Incision/Superficial (>30d post implant) (Infections and infestations) | 2
Suspected infection Incisional/Superficial (= 30d post implant) (Infections and infestations) | 10
Suture revision (Skin and subcutaneous tissue disorders) | 1
Syncope related to VT/VF Subject (Cardiac disorders) | 1
Systemic infection (Infections and infestations) | 1
T-wave oversensing (Product Issues) | 1
Transient Ischemic Attack (TIA) (Vascular disorders) | 1
Unable to convert VT/VF with S-ICD (Injury, poisoning and procedural complications) | 2
User error programmer (Product Issues) | 1
VT/VF below programming rate (Cardiac disorders) | 1
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 6
Vomiting during anesthesia induction (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study endpoints are compared against a performance goal rather than to a randomized control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02433379/Prot_SAP_000.pdf